CLINICAL TRIAL: NCT02468141
Title: Effect of Sipjeondaebo-tang for Cancer Related Anorexia in Cancer Patients: A Randomized Double Blinded Placebo Controlled Pilot Study
Brief Title: Effect of Sipjeondaebo-tang for Cancer Related Anorexia in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Gyu Ko, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KCRD_SJDBT_2015
Record Dates: First submitted 2015-05-27; First posted 2015-06-10 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cancer-related Problem/Condition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SJDBT group (Experimental): Herbal medicine
  Interventions: Drug: SJDBT
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SJDBT — Sipjeondaebo-tang
  Other Names: Sipjeondaebotang
  Arms: SJDBT group
Drug: Placebo — Placebo
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
To determine efficacy and safety of Sipjeondaebo-tang for Cancer patients suffering from anorexia after chemotherapy. Sipjeondaebo-tang will be administered for 4 weeks, 3 times per day after a meal. Changes of FAACT scale, Anorexia VAS, Weight, BMI, Clinical laboratory test such as ACTH, Cortisol, Chrelin, IL-6, ESR, CRP will be measured and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 20 to 80 years
* Individuals who are suffering from cancer-associated anorexia
* Patients within 1 month after completion of chemotherapy
* No plan for additional chemotherapy or radiotherapy
* Anorexia visual analogue scale (VAS) ≥ 40/100mm
* Qi deficiency scale ≥ 30 or Blood deficiency scale ≥ 30
* Neutrophil ≥ 1,500/㎕, platelet ≥ 100,000/㎕
* Total bilirubin lower than upper limit of normal (1.2 mg/㎗)
* ALT, AST lower than 2-fold the upper limit of normal
* Creatinine lower than 1.5 fold the upper limit of normal(1.09 mg/㎗)
* Written informed consent for participation in the trial

Exclusion Criteria:

* Patient impossible to oral intake
* Patient 5 years after cancer diagnosis
* ECOG performance status score > 3
* Patient with dementia, delirium, depression
* Patient who complain of more than 7 points when we use Numeric Rating Scale, which can affect appetite or calorie intake, within 2 weeks of screening
* Patient with diseases which can influence on appetite (such as hypoadrenalism, etc)
* Patient who are taking appetizers (such as megestrol acetate, corticosteroids, thalidomide)
* Women who has possibility of a pregnancy
* Others who are judged not to be appropriate to study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The Functional Assessment of Anorexia/Cachexia Therapy - Anorexia Cachexia Subscale | 4 weeks
  Function scores as measured by the likert scale

SECONDARY OUTCOMES:
FAACT scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chunhoo Cheon, Master, Study Director — Institute of Safety and Efficiency Evaluation for Korean Medicine
Locations (1):
- Dunsan Korean Medicine Hospital, Daejeon, South Korea

REFERENCES:
- [Derived] Cheon C, Yoo JE, Yoo HS, Cho CK, Kang S, Kim M, Jang BH, Shin YC, Ko SG. Efficacy and Safety of Sipjeondaebo-Tang for Anorexia in Patients with Cancer: A Pilot, Randomized, Double-Blind, Placebo-Controlled Trial. Evid Based Complement Alternat Med. 2017;2017:8780325. doi: 10.1155/2017/8780325. Epub 2017 Dec 26. PMID 29441116
- [Derived] Cheon C, Park S, Park YL, Huang CW, Ko Y, Jang BH, Shin YC, Ko SG. Sipjeondaebo-tang in patients with cancer with anorexia: a protocol for a pilot, randomised, controlled trial. BMJ Open. 2016 May 12;6(5):e011212. doi: 10.1136/bmjopen-2016-011212. PMID 27173813